CLINICAL TRIAL: NCT00657956
Title: Prospective RCT Using Roentgen Stereophotogrammetric Analysis (RSA) to Evaluate Fixation of the Biofoam Advance Total Knee Arthroplasty Components With and Without Screw Augmentation
Brief Title: Roentgen Stereophotogrammetric Analysis (RSA) to Evaluate Fixation of Biofoam Advance Total Knee Arthroplasty Components
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Principal Investigator, Michael Dunbar, MD, PhD, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dal07-02; CDHA-RS/2007-250 (Other: Capital District Health Authority Halifax Nova Scotia)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; arthroplasty; knee joint; radiography; surgery; Bone Density; Outcome Assessment (Health Care)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Advance Biofoam porous metal backed tibial component with or without screw augmentation — total knee arthroplasty tibial component that has a backing of porous titanium metal to facilitate bone in-growth

SUMMARY:
Hip and knee replacement arthroplasty are profoundly successful operative interventions, however, some joint replacements do fail and the life expectancy of a hip or knee arthroplasty is finite. This fact has largely been responsible for the continued development of new devices and techniques for joint arthroplasty surgery. Unfortunately, the introduction of new technologies and devices is not a benign process, and even subtle changes to existing implants can have a disastrous effect on patient outcome. The fact that new technologies and devices can lead to poor results has led some authors to advocate a phased introduction of new technologies. A key component of the phased introduction approach advocates the use of roentgen stereophotogrammetric analysis (RSA) early in the testing process. RSA is a highly accurate radiographic technique developed in Lund, Sweden and has for some time been the gold standard in Europe for assessing the stability of implants within bone. The purpose of this study is to utilize RSA to elucidate the migration patterns of the foam metal backed Advance Knee Arthroplasty components during the first 2 years postoperatively and to determine in what proportion of cases adequate fixation is achieved. In addition outcome measures will be recorded to quantify changes in functional status of subjects after surgery and bone mineral density will be monitored to quantify bone in-growth around the implant. Migration patterns will be compared to results obtained from previous studies of uncemented and cemented total knee arthroplasty components conducted at this centre.

DETAILED DESCRIPTION:
Hip and knee replacement arthroplasty are profoundly successful operative interventions, however, some joint replacements do fail and the life expectancy of a hip or knee arthroplasty is finite. This fact has largely been responsible for the continued development of new devices and techniques for joint arthroplasty surgery. Unfortunately, the introduction of new technologies and devices is not a benign process, and even subtle changes to existing implants can have a disastrous effect on patient outcome.

The fact that new technologies and devices can lead to poor results has led some authors to advocate a phased introduction of new technologies. A key component of the phased introduction approach advocates the use of roentgen stereophotogrammetric analysis (RSA) early in the testing process.

RSA is a highly accurate radiographic technique developed in Lund, Sweden and has for some time been the gold standard in Europe for assessing the stability of implants within bone. It is at least ten times more accurate than conventional radiography. RSA involves the insertion of small tantalum markers (0.8mm) into the bone and prosthesis at the time of surgery. By using a calibrated cage with additional markers and simultaneous bi-planar x-rays, micromotion at the prosthesis-bone interface can be very precisely determined. Two types of micromotion can be investigated: migration, i.e. gradual motion over time, and inducible displacement, i.e. instant motion in response to external forces. The pattern of micromotion exhibited by various prostheses and fixation techniques within the first post-operative year has been shown to be predictive of the long-term fixation of the component to bone, especially when considering the tibial prosthesis-bone interface. The value of this precise radiographic technique is that new technologies and techniques can be introduced in vivo while limiting their exposure to as few patients as possible. RSA is a proven, safe and invaluable method for assessing methods of knee component fixation as well as different design concepts.

DEXA bone densitometry has been demonstrated as a reliable method for determination bone mineral density about knee and hip implants. This technique provides further detail about the quality of fixation of knee and hip prostheses and implant induced bone remodeling.

The foam metal backed Advance Knee Arthroplasty components utilize a porous titanium coating on the non-articulating surface of the components to enhance the implant-bone interface. This 3-dimensional scaffold should promote bone in-growth that may provide a more robust bone-implant interface. The high coefficient of friction provides initial fixation negating the need for bone cement which should reduce duration of surgery. There is also a version of the Biofoam Advance that incorporates screwed fixation that allows for augmented fixation with up to four titanium screws, however, it is not clear that this augmentation is necessary.

The implant is based on previous proven designs from Wright Medical such as the Whiteside and Advance Medial Pivot. It incorporates the polyethylene, tibial tray and stem design from the Advance Medial Pivot and four stabilizing pegs on the underside of the tibial component that were used in the Whiteside. Of particular interest is the modularity of the Biofoam design, both the polyethylene and the tibial stem are attached to the tibial tray intraoperatively with the stem held in place with a morse taper, potentially providing the surgeon more sizing and positioning options during surgery.

Study Objective The purpose of this study is to utilize RSA to elucidate the migration patterns of the foam metal backed Advance Knee Arthroplasty components during the first 2 years postoperatively and to determine in what proportion of cases adequate fixation is achieved. In addition outcome measures will be recorded to quantify changes in functional status of subjects after surgery and bone mineral density will be monitored to quantify bone in-growth around the implant. Migration patterns will be compared to results obtained from previous studies of uncemented and cemented total knee arthroplasty components conducted at this centre.

Study Design This is a consecutive sample randomized control trial of patients undergoing total knee arthroplasty with the foam metal backed Advance Biofoam Knee Arthroplasty system (Wright Medical Inc.) with and without screws utilizing RSA to identify the migration patterns of the tibial and femoral components of the implant. DEXA scanning will also be conducted to determine changes in the bone mineral density adjacent to the implant. Health status and functional outcome measures will be recorded to quantify functional status of subjects before surgery and at each follow-up interval.

Statement of research questions Question 1: Is there a difference in fixation to the proximal tibia between tibial components fixed with screws and those without screws?

Null Hypothesis:

There is no significant difference in micromotion patterns of the foam metal backed arthroplasty components fixed with screws and those fixed without.

Alternative Hypothesis:

There are significant differences in micromotion patterns between the tibial components fixed with screws and those fixed without.

Question 2: Do the screwed components achieve adequate fixation to the underlying bone?

Null Hypothesis:

There is no significant continuous migration at 2 years with the screwed components indicating adequate long-term fixation at the implant - bone interface.

Alternative Hypothesis:

There is significant continuous migration at 2 years with the screwed components indicating inadequate fixation at the implant - bone interface.

Question 3: Do the unscrewed components achieve adequate fixation to the underlying bone?

Null Hypothesis:

There is no significant continuous migration at 2 years with the unscrewed components indicating adequate long-term fixation at the implant - bone interface.

Alternative Hypothesis: There is significant continuous migration at 2 years with the unscrewed components indicating inadequate fixation at the implant - bone interface.

Question 4: What are the migration patterns (translations and rotations) of the foam metal backed arthroplasty components during the first two years postoperatively and how do they compare between those fixed with screws and those fixed without screws?

Question 5: For what proportion of implants in each group does migration continue to increase during the two year follow-up?

Question 6: Is there a significant difference in health status and functional outcome before and after total knee arthroplasty using foam metal backed arthroplasty components?

Question 7: Are there significant difference in bone mineral density between the operative knee (distal femur and proximal tibia) and other body sites over time?

Subjects n= 21 per group

Allowing for 20% lost to follow-up a total sample size of 50 (25 per group) will be sufficient to elucidate a significant difference in micromotion (clinically significant motion defined as ≥ 0.2 mm) between groups.

Subjects will be screened consecutively and enrolled from clinic after informed consent has been obtained. Their vital information and co-morbidities will be recorded from the chart and functional status will be assessed using the KSCRS, SF-36, WOMAC, Oxford 12 knee score, UCLA Activity Level, Self-Administered Comorbidity Questionnaire (SCQ), the Pain and Catastrophizing Scale (PCS) and visual analogue scales for pain and health status. All information will be kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating surgical intervention
* Between the ages of 21 and 80 inclusive
* Ability to give informed consent

Exclusion Criteria:

* Significant co-morbidity affecting ability to ambulate
* Flexion contracture greater than 15°
* Extension lag greater than 10°
* Tibial subluxation greater than 10 mm on standing AP radiograph
* Prior arthroplasty, patellectomy or osteotomy with the affected knee
* Lateral or medial collateral ligament instability (> 10° varus/valgus)
* Leg length discrepancy greater than 10 mm
* Active or prior infection
* Morbid Obesity (BMI > 40)
* Medical condition precluding major surgery
* Severe osteoporosis or osteopenia
* Neuromuscular impairment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
micromotion of tibial component as measured with RSA | 2 years postoperative

SECONDARY OUTCOMES:
Bone mineral density around the tibial component | 2 years postoperative
Subjective health outcome questionnaires - SF36, WOMAC, Oxford12 knee, Pain and Catastrophizing Scale, Standardized comorbidity questionnaire | 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gross, MD, Principal Investigator — Dalhousie University; Michael J Dunbar, MD PhD, Study Director — Dalhousie University
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada